CLINICAL TRIAL: NCT01293396
Title: Comparison of the Impact of Biphasic Insulin Aspart 30 (BiAsp 30), Biphasic Insulin Aspart 70 (BiAsp 70) and Insulin Aspart on Postprandial Glucose and Lipid Metabolism During Two Consecutive Meals in Type 2 Diabetics.
Brief Title: Comparison of Premixed Insulins Aspart 30, Aspart 70 and Aspart on Postprandial Lipids
Acronym: HUCKEPACK2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ENM-DA-008; 2008-008486-35 (EudraCT Number)
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes
Keywords: insulin aspart 30; insulin aspart 70; insulin aspart; postprandial glucose and lipid metabolism; consecutive mixed meals
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biphasic Insulin Aspart 30 (Active Comparator): 35% of their usual total daily insulin dose before the standardized breakfast and 25% prior to lunch
  Interventions: Drug: Insulin Aspart 30
- Biphasic Insulin Aspart 70 (Active Comparator): 35% of their usual total daily insulin dose before the standardized breakfast and 25% prior to lunch
  Interventions: Drug: Insulin Aspart 70
- Insulin Aspart (Active Comparator): 35% of their usual total daily insulin dose before the standardized breakfast and 25% prior to lunch
  Interventions: Drug: Insulin Aspart

INTERVENTIONS:
Drug: Insulin Aspart — Patients received insulin aspart before breakfast and before lunch.
  Other Names: Novorapid
  Arms: Insulin Aspart
Drug: Insulin Aspart 30 — Patients received biphasic insulin aspart 30 before breakfast and before lunch.
  Other Names: Novomix 30
  Arms: Biphasic Insulin Aspart 30
Drug: Insulin Aspart 70 — Patients received biphasic insulin aspart 70 before breakfast and before lunch.
  Other Names: Novomix 70
  Arms: Biphasic Insulin Aspart 70

SUMMARY:
The aim of the study is to investigate meal-related treatment with either premixed Insulin Aspart 30, Aspart 70 and Aspart with regard to postprandial glucose, triglyceride and free fatty acids excursions after a standard breakfast and lunch.

DETAILED DESCRIPTION:
Whereas the effects of each of the established types of insulin (remixed Insulin Aspart 30, Aspart 70 and Aspart) have been shown before, their specific glucose and lipid lowering capacities have so far not been investigated in a simulated physiological situation.

ELIGIBILITY:
Inclusion Criteria:

* Type-II Diabetes
* BMI > 27 kg/m2
* age 35 to 75 years
* HbA1c < 8.5%
* informed consent
* treatment with pre-mixed insulin
* stabile dose of insulin for at least 4 weeks

Exclusion Criteria:

* Type-I Diabetes mellitus
* HbA1c > 8.5 %
* Serum Creatinine > 1.7 mg/dl
* Alaninaminotranferase or Aspartataminotransferase > 3x Upper Limit of Normal
* treatment with sulfonylurea or gliptins
* treatment with glitazones
* manifest clinical infections
* treatment with glucocorticoids or antipsychotic drugs
* psychiatric diseases
* alcohol abuse
* myocardial infarction or stroke within the previous 3 months
* surgery within the previous 3 months

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Sourij, MD, Principal Investigator — Medical University of Graz, 8036 Graz, Austria
Locations (1):
- Medical University of Graz, Department for Internal Medicine, Graz, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 patients were screened and in total 20 randomizations were performed. After randomization 20 randomized subjects finished all three study visits.
Pre-assignment Details: All subjects received all of the three insulins within various sequences in a randomized order. Randomisation lists for the insulin sequence were provided by a researcher otherwise not involved in the clinical trial performance.
Groups:
- Group 1; Group 2; Group 3: Participants were randomized to each intervention and re-randomized to the remaining interventions after each washout period.
Period: First Intervention
Arm/Group | Group 1 | Group 2 | Group 3
Started | 6 | 7 | 7
Completed | 6 | 7 | 7
Not Completed | 0 | 0 | 0
Period: Wash Out Period 1 (3 Days)
Arm/Group | Group 1 | Group 2 | Group 3
Started | 6 | 7 | 7
Completed | 6 | 7 | 7
Not Completed | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Group 1 | Group 2 | Group 3
Started (20 participants finished washout-period 1 and were randomized to the 3 interventions (BiAsp30, BiAsp70 and IAsp). In this cross over design the participants first received BiAsp30, then e.g. switched to BiAsp70 and then to IAsp. Therefore, the number of participants could not be the same to participants who completed previous period. However, the total number of partcipants who finished the washout period is equal to the number of particpants who started this intervention sequence.) | 5 | 5 | 10
Completed | 5 | 5 | 10
Not Completed | 0 | 0 | 0
Period: Wash Out Period 2 (3 Days)
Arm/Group | Group 1 | Group 2 | Group 3
Started | 5 | 5 | 10
Completed | 5 | 5 | 10
Not Completed | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Group 1 | Group 2 | Group 3
Started (20 participants finished washout-period 2 and were randomized to the 3 interventions (BiAsp30, BiAsp70 and IAsp).) | 9 | 8 | 3
Completed | 9 | 8 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: 20 patients with type 2 diabetes receive insulin aspart, premixed biphasic insulin 30 and premixed biphasic insulin aspart 70 in randomized order.
Arm/Group | Overall Study
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (6)
Sex: Female, Male [Count of Participants; unit: Participants] — Measure Type: Count of Participants Unit of measure: participants
  Participants
    Female | 6
    Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Over Basal for Postprandial Glucose From 0 to 600min
Description: Area over basal for postprandial glucose from 0 (Fasting glucose, measured at daily study start) to 600 min (after breakfast) Area over basal is calculated according to the trapezoidal rule.
Time Frame: 0,30,60,90,120,180,240,270,300,330,360,420,480,540,600 minutes post-dose (daily study start)
Measure: Mean (Standard Deviation); unit: mg*/min/dL
Arm/Group | Biphasic Insulin Aspart 30 | Biphasic Insulin Aspart 70 | Insulin Aspart
Number analyzed (Participants) | 20 | 20 | 20
mg*/min/dL | 591 (681) | 220 (617) | 197 (550)

2. Primary Outcome: Area Over Basal for Postprandial Triglycerides
Description: Area over basal for postprandial triglycerides from 0 (Fasting triglycerides, measured at daily study start) to 600 min (after breakfast) Area over basal is calculated according to the trapezoidal rule.
Time Frame: 0,30,60,90,120,180,240,270,300,330,360,420,480,540,600 minutes post-dose (daily study start)
Measure: Mean (Standard Deviation); unit: mg*min/dL
Arm/Group | Biphasic Insulin Aspart 30 | Biphasic Insulin Aspart 70 | Insulin Aspart
Number analyzed (Participants) | 20 | 20 | 20
mg*min/dL | 484 (342) | 358 (544) | 412 (831)

3. Secondary Outcome: Maximum Glucose Increase
Description: Maximum glucose increase from baseline to 600min after baseline
Time Frame: 0,30,60,90,120,180,240,270,300,330,360,420,480,540,600 minutes post-dose (daily study start)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Biphasic Insulin Aspart 30 | Biphasic Insulin Aspart 70 | Insulin Aspart
Number analyzed (Participants) | 20 | 20 | 20
mg/dL | 89.25 (57.85) | 55.95 (42.44) | 60.25 (40.45)

4. Secondary Outcome: Maximum Triglyceride Increase
Description: Maximum trigylceride increase from Baseline to 600min after Baseline
Time Frame: 0,30,60,90,120,180,240,270,300,330,360,420,480,540,600 minutes post-dose (daily study start)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Biphasic Insulin Aspart 30 | Biphasic Insulin Aspart 70 | Insulin Aspart
Number analyzed (Participants) | 20 | 20 | 20
mg/dL | 484 (342) | 358 (544) | 412 (831)

5. Secondary Outcome: Area Over Basal for Postprandial Insulin
Description: Area over basal for postprandial insulin from 0 (Fasting insulin, measured at daily study start) to 600 min (after breakfast) Area over basal is calculated according to the trapezoidal rule.
Time Frame: 0,30,60,90,120,180,240,270,300,330,360,420,480,540,600 minutes post-dose (daily study start)
Measure: Mean (Standard Deviation); unit: µU*min/L
Arm/Group | Biphasic Insulin Aspart 30 | Biphasic Insulin Aspart 70 | Insulin Aspart
Number analyzed (Participants) | 20 | 20 | 20
µU*min/L | 211.2 (149.7) | 141.2 (155.3) | 128.6 (106.7)

6. Secondary Outcome: Area Over Basal for Postprandial C-peptide
Description: Area over basal for postprandial c-peptide from 0 (Fasting c-peptide, measured at daily study start) to 600 min (after breakfast) Area over basal is calculated according to the trapezoidal rule.
Time Frame: 0,30,60,90,120,180,240,270,300,330,360,420,480,540,600 minutes post-dose (daily study start)
Measure: Mean (Standard Deviation); unit: mg*min/mL
Arm/Group | Biphasic Insulin Aspart 30 | Biphasic Insulin Aspart 70 | Insulin Aspart
Number analyzed (Participants) | 20 | 20 | 20
mg*min/mL | 21.6 (14.1) | 12.8 (11.5) | 13.4 (11.8)

ADVERSE EVENTS:
Arm/Group | Biphasic Insulin Aspart 30 | Biphasic Insulin Aspart 70 | Insulin Aspart
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 2/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biphasic Insulin Aspart 30 (N=20) | Biphasic Insulin Aspart 70 (N=20) | Insulin Aspart (N=20)
Mild Hypoglycaemic Event (Endocrine disorders) | 1 (2) | 2 (4) | 2 (2) — Hypoglycaemic events blood glucose levels <70mg/dL
Moderate Hypoglycaemic Event (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) — Hypogylcaemic Event <54mg/dL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes